CLINICAL TRIAL: NCT04279769
Title: A Phase 1b Randomized, Double-blind, Placebo-Controlled Trial to Evaluate the Safety of CB-280 in Patients With Cystic Fibrosis
Brief Title: Study to Evaluate the Safety of CB-280 in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CX-280-202
Record Dates: First submitted 2020-02-10; First posted 2020-02-21 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Cystic Fibrosis
Keywords: Arginase inhibitor; CB-280
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): CB-280 twice daily at 50 mg for 14 days
  Interventions: Drug: CB-280
- Cohort 2 (Experimental): CB-280 twice daily at 100 mg for 14 days
  Interventions: Drug: CB-280
- Cohort 3 (Experimental): CB-280 twice daily at 200 mg for 14 days
  Interventions: Drug: CB-280
- Cohort 4 (Experimental): CB-280 twice daily at 400 mg for 14 days
  Interventions: Drug: CB-280
- Placebo (Placebo Comparator): Placebo twice daily for 14 days
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: CB-280 — CB-280, oral capsule administered twice daily at the assigned dose level for 14 days
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4
Drug: Placebos — Placebo oral capsule administrated twice daily at the assigned dose level for 14 days
  Arms: Placebo

SUMMARY:
This is a phase 1b multiple ascending dose escalation study to evaluate the safety and tolerability of arginase inhibitor CB-280 in subjects with cystic fibrosis.

DETAILED DESCRIPTION:
Study CX-280-202 is a Phase 1b, randomized, double-blind, placebo-controlled, multiple ascending dose escalation study of CB-280 in adult subjects with cystic fibrosis and chronic infection with Pseudomonas aeruginosa. The study will evaluate the safety, pharmacokinetics, pharmacodynamics, and biological activity of CB-280 in approximately 32 adult patients with cystic fibrosis. There are four planned sequential dose escalation cohorts of 8 subjects each, randomized 6:2 to receive CB-280 or matched placebo at doses of 50 mg, 100 mg, 200 mg, or 400 mg administered twice daily for 14 days. Intermediate dose levels may be evaluated based on emerging safety data at the planned dose levels.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent in accordance with federal, local, and institutional guidelines
2. Confirmed diagnosis of cystic fibrosis
3. Male or female subjects ≥ 18 years on the date of informed consent
4. Percent predicted FEV1 of 40-90% at screening per Global Lung Function Initiative (GLI) equation
5. Clinically stable with no significant changes in health status within 28 days prior to Day 1
6. Chronic lung infection with P. aeruginosa defined as at least one positive culture in the last two years and more than 50% of cultures positive since then
7. Stable cystic fibrosis medication regimen for at least 28 days inclusive of CFTR modulators prior to Day 1
8. Hemoglobin > 10 g/dL at screening
9. Glomerular filtration rate > 50 mL/min/1.73 m2 at screening
10. Normal liver function at screening

Exclusion Criteria:

1. History of any comorbidity that, in the opinion of the Investigator, might pose an additional risk in administering study drug to the subject or confound the results of the study
2. Lung infection with organisms associated with a more rapid decline in pulmonary status (including, but not limited to, Burkholderia cenocepacia, Burkholderia dolosa, and Mycobacterium abscessus)
3. Unable to receive study medication per os (PO)
4. Females who are pregnant, have a positive pregnancy test at screening, or are nursing (lactating)

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Determine the safety and tolerability of CB-280 in adult cystic fibrosis patients: incidence and severity of adverse event (AEs) assessed by Common Terminology Criteria for Adverse Events, version 5 (CTCAE v5.0) | Start of treatment to Day 28

SECONDARY OUTCOMES:
Pharmacokinetics of plasma CB-280 measured by Peak Plasma Concentration (Cmax) | Day 14
Pharmacokinetics of plasma CB-280 measured by area under the plasma concentration versus time curve, from time 0 to the last observed non-zero concentration (AUC 0-t) | Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Emil T Kuriakose, MD, Study Director — Calithera Bioscience
Locations (20):
- United States (17):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Long Beach Memorial Medical Center, Long Beach, California
  - University of Florida, Gainesville, Florida
  - The Cystic Fibrosis Institute, Glenview, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Brigham & Women's Hospital, Boston, Massachusetts
  - Billings Clinic, Billings, Montana
  - New York Medical College at Westchester Medical Center, Hawthorne, New York
  - UNC Marsico Clinical Research Center, Chapel Hill, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Hershey Medical Center Pennsylvania State University, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Utah, Salt Lake City, Utah
  - Vermont Lung Center at the University of Vermont Medical Center, Colchester, Vermont
  - Virginia Commonwealth University, Richmond, Virginia
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - St. Pauls' Hospital, Vancouver, British Columbia
  - McGill University Health Center, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No